CLINICAL TRIAL: NCT02983630
Title: Allergy Testing of Primary Care Patients Labeled as Penicillin Allergic
Brief Title: Allergy Testing of Patients Labeled as Penicillin Allergic
Status: Completed | Type: Observational
Sponsor: Albany Medical College (Other)
Responsible Party: Principal Investigator, Britta Sundquist, Instructor of Medicine, Albany Medical College
Other Study IDs: 4479
Record Dates: First submitted 2016-09-22; First posted 2016-12-06 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Drug Hypersensitivity
MeSH Terms: conditions — Drug Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Penicillin allergy testing — The standard protocol for testing for penicillin hypersensitivity, including initial skin testing with prick and intradermal evaluation followed by oral challenge if skin testing is negative.

SUMMARY:
Patients labeled as penicillin allergic, rarely have this confirmed and being labeled as "penicillin allergic" is associated with increased health care costs, adverse effects and antibiotic resistance. The investigators will recruit participants from primary care practices labeled as penicillin allergic and offer allergy testing. The aim of this study is to develop a community, outpatient program for evaluation of penicillin allergy.

ELIGIBILITY:
Inclusion Criteria:

1. Labeled as having penicillin or amoxicillin allergy
2. Family history of penicillin allergy

Exclusion Criteria:

1. History of beta-lactam associated toxic epidermal necrolysis/Stevens Johnson syndrome to penicillin or amoxicillin
2. History of Drug induced Eosinophilia with Systemic Symptoms (DRESS)
3. History of drug induced: autoimmune hepatitis/interstitial nephritis, or hemolytic anemia
4. Poorly controlled asthma or heart disease
5. Currently pregnant
6. Unable to discontinue certain medications that may interfere with testing including (antihistamines, steroids, beta-blockers, tricyclic antidepressants, omalizumab)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults ages 18 and older from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Allergy testing for penicillin allergy results | 6 months

SECONDARY OUTCOMES:
Participant satisfaction after allergy testing with follow-up questionnaire | Within 6 months following testing
  A questionnaire will be provided to participants to review their experience with penicillin allergy testing, whether they will take penicillin in the future and if it is valuable information to be tested. Answers will be yes and no. This information will tell us
Development of new drug allergies following negative testing questionnaire | 6 months-2 years
  Follow-up questionnaire will be sent to participants to evaluate whether they have needed any antibiotics and if so, whether they've had any reactions. This will be two yes/no questions to assess the incidence of development of new allergic reaction following negative testing.

CONTACTS AND LOCATIONS:
Locations (1):
- Albany Medical College Allergy, Asthma and Immunology Center, Albany, New York, United States